CLINICAL TRIAL: NCT00002397
Title: An Exploratory Study of Fortovase (Saquinavir) Soft Gelatin Capsules (SGC) Plus d4T and 3TC or Fortovase (Saquinavir) SGC Plus Nelfinavir and d4T in Patients With HIV-1 Associated Nephropathy
Brief Title: A Study of Saquinavir Soft Gel Capsules (SGC) Used in Combination With Two Other Anti-HIV Drugs in Patients With HIV-Associated Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 229P; NR15690/M61021
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: HIV Infections; AIDS-Associated Nephropathy
Keywords: Kidney Failure, Chronic; HIV-1; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Lamivudine; Saquinavir; AIDS-Associated Nephropathy; Reverse Transcriptase Inhibitors; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections; AIDS-Associated Nephropathy; Kidney Failure, Chronic | interventions — Nelfinavir; Saquinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Saquinavir
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of saquinavir SGC plus stavudine (d4T) plus lamivudine (3TC) with that of saquinavir SGC plus nelfinavir plus d4T in patients with HIV-associated kidney disease. This study examines whether these drug combinations are effective in preventing kidney disease from progressing to a stage where it is immediately life threatening. This study also examines the effect these drug combinations have on the level of HIV detected in these patients. Finally, this study evaluates the drug level (the amount of drug found in the body) of these two combinations in patients with kidney disease.

DETAILED DESCRIPTION:
This is an open-label, non-comparative, randomized, single center, 24-week study. Patients are stratified into 3 groups (8 patients in each group) based on kidney function:

Group 1: Serum creatine less than 2 mg/dL. Group 2: Serum creatine 2-5 mg/dL. Group 3: Serum creatine greater than 5 mg/dL.

All 24 patients are randomized 1:1 to receive 1 of 2 study regimens:

Arm A: Saquinavir SGC plus d4T plus 3TC. Arm B: Saquinavir SGC plus nelfinavir plus d4T. Patients are seen at Weeks 4, 8, 12, and 24. At Week 24, a kidney biopsy is performed with patient consent.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Detectable HIV-1 RNA by Amplicor assay.
* Biopsy-proven nephropathy.

Exclusion Criteria

Prior Medication:

Excluded:

* Saquinavir and nelfinavir.
* d4T or 3TC within the past 4 months.

Required:

Stable antiretroviral therapy for more than 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Med Ctr, New York, New York, United States